CLINICAL TRIAL: NCT04156932
Title: Closure at the Origin of the Uterine Artery vs. Closure at the Cervico-isthmic Level in Laparoscopic Hysterectomy: a Randomized Clinical Trial
Brief Title: Closure of the Uterine Artery at Its Origin vs at the Cervix: a Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale degli Infermi di Biella (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 440/CE
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Anatomy; Laparoscopy; Uterine Artery; Hysterectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OUC (Active Comparator): Origin uterine artery closure
  Interventions: Procedure: uterine artery closure
- IUC (Active Comparator): Cervical-isthmic uterine artery closure
  Interventions: Procedure: uterine artery closure

INTERVENTIONS:
Procedure: uterine artery closure — Interruption the uterine blood flow by closing the uterine artery at its cervical-isthmic part or at its origin.

SUMMARY:
One of the fundamental surgical steps in patients undergoing laparoscopic hysterectomy is the closure of the uterine artery, this vessel provides the greatest blood supply to the uterus.

This step can be done in two ways: the surgeon can choose to interrupt the blood flow by closing the uterine artery in its last part, close to the uterus, or the surgeon can develop the anatomical spaces around the uterus into the deep pelvis, closing it to its origin, maintaining a minimally invasive approach in both cases.

Scientific research has tried to establish whether one of the two modalities is the best in reducing intraoperative blood loss and possible complications, but currently there is not enough evidence to recommend an approach rather than another.

The investigator has therefore decided to evaluate the results at the end of a laparoscopic hysterectomy in a scientifically rigorous manner.

ELIGIBILITY:
Inclusion Criteria:

* benign disease
* elective laparoscopic hysterectomy

Exclusion Criteria:

* malignant disease
* emergency laparoscopic hysterectomy

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
estimated blood loss | End of surgical procedure
  ml

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale degli Infermi, Ponderano, Biella, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aarts JW, Nieboer TE, Johnson N, Tavender E, Garry R, Mol BW, Kluivers KB. Surgical approach to hysterectomy for benign gynaecological disease. Cochrane Database Syst Rev. 2015 Aug 12;2015(8):CD003677. doi: 10.1002/14651858.CD003677.pub5. PMID 26264829
- [Result] Aust T, Reyftmann L, Rosen D, Cario G, Chou D. Anterior approach to laparoscopic uterine artery ligation. J Minim Invasive Gynecol. 2011 Nov-Dec;18(6):792-5. doi: 10.1016/j.jmig.2011.07.008. PMID 22024265
- [Result] Simpson NA, Nimrod C, De Vermette R, Leblanc C, Fournier J. Sonographic evaluation of intervillous flow in early pregnancy: use of echo-enhancement agents. Ultrasound Obstet Gynecol. 1998 Mar;11(3):204-8. doi: 10.1046/j.1469-0705.1998.11030204.x. PMID 9589145
- [Result] Uccella S, Cromi A, Casarin J, Bogani G, Serati M, Gisone B, Pinelli C, Fasola M, Ghezzi F. Minilaparoscopic versus standard laparoscopic hysterectomy for uteri >/= 16 weeks of gestation: surgical outcomes, postoperative quality of life, and cosmesis. J Laparoendosc Adv Surg Tech A. 2015 May;25(5):386-91. doi: 10.1089/lap.2014.0478. Epub 2015 Apr 3. PMID 25839384
- [Result] Uccella S, Cromi A, Serati M, Casarin J, Sturla D, Ghezzi F. Laparoscopic hysterectomy in case of uteri weighing >/=1 kilogram: a series of 71 cases and review of the literature. J Minim Invasive Gynecol. 2014 May-Jun;21(3):460-5. doi: 10.1016/j.jmig.2013.08.706. Epub 2013 Sep 4. PMID 24012921